CLINICAL TRIAL: NCT03733509
Title: Intraoperative Direct Adductor Canal Nerve Block Versus Post Operative Ultrasound Guided Adductor Canal Nerve Block in Total Knee Arthroplasty: a Double-blind Randomized Trial
Brief Title: Intraoperative Direct vs Postoperative Ultrasound Guided Adductor Canal Nerve Block After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 180620002
Record Dates: First submitted 2018-11-06; First posted 2018-11-07 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Knee Osteoarthritis; Total Knee Arthroplasty; Nerve Block
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Two arm, randomly assigned
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Total blind (patient, physicians, outcome assessors and statistician) Closed envelope by independent randomizer is given to physician assistant. The assistant prepares randomly allocated placebo or local anesthetic. Group is coded so that statistician is also blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraoperative Block (Experimental): Before skin closure, blunt suprapatellar dissection proximal to medial femoral condyle towards adductor canal. Nerve block at this level with 20ml of Bupivacaine 0.25%.
  Postoperatively, mid-thigh ultrasound guided standard adductor canal nerve block with 20ml of saline solution (NaCl 0.9%).
  Interventions: Procedure: Intraoperative Block; Procedure: Ultrasound Placebo
- Ultrasound Block (Active Comparator): Before skin closure, blunt suprapatellar dissection proximal to medial femoral condyle towards adductor canal. Nerve block at this level with 20ml of of saline solution (NaCl 0.9%).
  Postoperatively, mid-thigh ultrasound guided standard adductor canal nerve block with 20ml Bupivacaine 0.25%.
  Interventions: Procedure: Ultrasound Block; Procedure: Intraoperative Placebo

INTERVENTIONS:
Procedure: Intraoperative Block — One shot adductor canal nerve block with 20ml of bupivacaine 0.25% through surgical incision
  Arms: Intraoperative Block
Procedure: Ultrasound Block — One shot adductor canal nerve block with 20ml of bupivacaine 0.25% mid-thigh
  Arms: Ultrasound Block
Procedure: Intraoperative Placebo — One shot adductor canal nerve infusion with 20ml of saline solution through surgical incision
  Arms: Ultrasound Block
Procedure: Ultrasound Placebo — One shot adductor canal nerve infusion with 20ml of saline solution mid-thigh
  Arms: Intraoperative Block

SUMMARY:
This study compares analgesic effect between two techniques of adductor canal nerve block after total knee arthroplasty. The first group of the patients will receive intraoperative adductor canal nerve block; and the other group post operative ultrasound guided adductor canal nerve block. Investigators will measure postoperative opioid consumption, pain management and rehabilitation goals.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is a successful alternative to treat late stage knee osteoarthritis (OA). Pain management has been one of the main focuses of postoperative care. Most surgeons prefer a comprehensive multimodal approach including preoperative pharmacological treatment, intraoperative infiltration with complex drug mixes and postoperative peripheral nerve block.

The most common postoperative nerve block alternative is the proximal femoral nerve block (FNB) which has shown improvements on postoperative pain measured by reduced opioid consumption and decreased pain at rest. Its main detractors argue that the motor nerve block effect is deleterious to early ambulation and have promoted adductor canal nerve blocks (ACB). Described by Lund et al in 2011, ACB block main femoral pain sensory contributors to the knee (articular branches of obturator nerve, vastus medialis branch and saphenous nerve) but is more distal to most motor branches to the quadriceps allowing near to normal quadriceps strength.

Standard ACB block is performed under ultrasound guidance after surgery completion, still in the operating room (OR). Recent literature has shown the anatomic feasibility of intraoperative ACB via blunt suprapatellar dissection in standard medial parapatellar TKA approaches. The study seeks to determine the effectiveness of standard ultrasound guidance ACB compared with intraoperative ACB.

ELIGIBILITY:
Inclusion Criteria:

* Primary total knee arthroplasty
* Unilateral
* American Society of Anesthesiologists (ASA) score I, II or III
* Accepts spinal anesthesia

Exclusion Criteria:

* General anesthesia
* Chronic kidney disease
* Drug or alcohol abuse
* Chronic opioid use
* Allergic to bupivacaine or similar

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
24 hour opioid consumption | First 24 hours after surgery
  Opioid consumption by patient controlled analgesia (PCA) and any other oral or IV analgesics

SECONDARY OUTCOMES:
24 patient reported pain | First 24 hours after surgery
  Patient reported pain scale using visual analog scale (VAS) every 6 hours after surgery (0 hours, 6 hours, 12 hours, 18 hours and 24 hours)
Time up and go Test | 24 hours after surgery
  Standardised test to determine patients ability to walk 24 hours after surgery
Time to Discharge | 7 days
  Time between surgery and patient in conditions for discharge: no IV requirements, basic walking capability and VAS pain score equal or below 3
Range of motion | 24 hours after surgery
  Active and passive knee range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Besa, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided